CLINICAL TRIAL: NCT00292136
Title: Real Time Assessment of Drug Craving, Use, and Abstinence During Outpatient: A Development and Feasibility Study
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999903385; 03-DA-N385
Record Dates: First submitted 2006-02-14; First posted 2006-02-15 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2013-06-11

CONDITIONS: Cocaine Addiction; Opiate Addiction
Keywords: Cocaine Dependence; Drug Relapse; Pharmacokinetics; EMA; Polydrug Abuse
MeSH Terms: conditions — Cocaine-Related Disorders; Opioid-Related Disorders

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

* The treatment of addiction often hinges on preventing relapse into drug-using behaviors, which occurs at high rates even after prolonged abstinence. Research has shown that constant reporting through personal data-collection devices, such as electronic diaries, can help prevent relapse and reinforce abstinence. This constant reporting is known as Ecological Momentary Assessment (EMA).
* The researchers here at NIDA have already completed two major arms of the study, focusing on patterns of craving and drug use during methadone maintenance, and on whether electronic diaries could help remind outpatients to complete treatment tasks. An ongoing arm of the study is examining connections among drug craving/use, stress, and geographical location.

Objective:

- To investigate the role of stress associated with geographical location in drug craving and use.

Eligibility:

- Individuals between 18 and 65 years of age or older who are dependent on opioids (cocaine and/or heroin).

Design:

* The study will last 28 weeks. After the initial screening, participants will receive daily methadone and weekly drug counseling sessions that will continue throughout the study.
* After 3 weeks of methadone treatment, participants will have 15 weeks of EMA in which they will record both event-triggered cravings and daily responses (3 per day). EMA will consist of event-triggered recordings (initiated by participants whenever they use heroin or cocaine, or whenever they feel an urge to do so) and random-signal-triggered recordings (3 per day). During EMA, participants will begin a voucher-based program to encourage abstinence from heroin and cocaine.
* Participants will also carry global positioning system (GPS) units to record their locations during these 15 weeks, and will complete questionnaires about stress levels at specific intervals during the study.
* At the end of the study, participants will have the choice of transferring to a community clinic or undergoing an 8-week taper from methadone.

DETAILED DESCRIPTION:
Background. We have already completed the original, major arm of this protocol (a natural-history study of craving and lapse). Still open for enrollment is the second minor arm (a within-subject trial of PDA-based treatment-task reminders). In the third arm there will be enhanced assessment of mood, stress, and geographical location to further study craving and lapse. All arms of the study have developed from either or both of two aspects of the original arm: (1) Our growing appreciation of the technical possibilities of electronic data collection in participants daily environments, and (2) our growing interest in having participants provide descriptive data about the day-to-day experience of addiction and recovery.

The major completed arm of the protocol has provided a wealth of descriptive data on drug craving and lapse via Ecological Momentary Assessment (EMA), in which participants carry handheld data-collection devices (electronic diaries, EDs) on which they report, in real time, their activities and moods. Beyond data monitoring, EDs can be used to complement behavioral interventions. The data-collection devices can be additionally programmed to prompt completion of therapist-assigned homework exercises; by extending support outside the therapy session, clinical outcome may be improved. Furthermore, there is an evidenced association between completion of homework exercises and therapeutic outcome. Adapting existing homework assignments to make them more engaging may increase homework completion and, in turn, general compliance with therapy (Arm 2). The rationale for the third arm of the study is to broaden the perspective of the examination of the natural history of drug cravings and lapses by refining our assessments of geographical location and the stressors associated with it. In doing so, we intend to investigate determinants of addiction that are not reducible to individual-level traits but are instead reflective of broader socioeconomic problems manifested in differences among neighborhoods.

Scientific goals. Arm 1) To investigate the relationships between putative triggers and drug craving and lapse; Arm 2) To investigate interactive effects of electronic-diary reminders, and simplified therapy-assigned homework tasks, on homework completion and therapeutic outcome; Arm 3) Using refinements in our assessment methods, to investigate the role of stress associated with geographical location in drug craving and use.

Participant population. Arm 2: 35 cocaine-abusing opioid-dependent outpatients. Arm 3: 50 cocaine-abusing opioid-dependent outpatients (separate from those in Arm 2). Target enrollment for both arms will include 40% women and 60% minorities (mostly African-American).

<TAB>

Experimental design and methods. After 3 weeks of stabilization on daily methadone, outpatients will undergo 25 weeks of EMA. EMA will consist of event-triggered recordings (initiated by participants whenever they use heroin or cocaine, or whenever they feel an urge to do so) and random-signal-triggered recordings (3 per day). Target quit dates for heroin and cocaine will occur, respectively, on the first and third weeks of EMA. Two days after the cocaine quit date, all participants will begin 12 weeks of intensive voucher-based contingency management to reinforce abstinence from heroin and cocaine. Arm 2: During the same 12 weeks, a within-subjects manipulation will occur: participants will receive simplified versions of the current counselor-assigned homework tasks, and participants will receive a daily reminder via the PDA to complete their homework tasks (whether they are standard or simplified versions). The simplified homework tasks and reminders will be given during two separate, counterbalanced, three-week blocks. Arm 3: Starting at week 4 and continuing through week 18 participants will answer enhanced EMA questions regarding stress, mood, location, drug craving and use. Additionally, participants in Arm 3 will carry GPS units to record their locations during these 15 weeks. GPS location will be examined with their drug use, craving and self-reported mood. They will also complete retrospective stress questionnaires at week 3 and then at 4-week intervals throughout the completion of the study: week 7, 11, 15, 19, 23, and 27. After the 12-week homework (Arm 2) or enhanced EMA phase (Arm 3) ends, participants will have the choice of transferring to a community clinic or undergoing an eight-week taper from methadone. For participants in Arm 2 who choose to detox at Archway, EMA may continue. However, for participants in Arm 3, no EMA or GPS data will be collected during the pre-detox or detox phase (weeks 19-28).

<TAB>

Benefits to participants and/or society. Direct benefits to participants include psychological and pharmacologic assistance for decreasing illicit drug use. The methadone administered during the study will decrease the participants intravenous opiate use. The contingency management and psychotherapy procedures may further reduce drug use and HIV risk behaviors. The decrease in HIV risk behaviors should result in lower incidence of HIV disease. Benefits to society include an increase in scientific understanding of the precipitants and process of craving, lapse, and relapse, and an improvement in our ability to assess the clinical effectiveness of relapse-prevention medications in future clinical trials.

<TAB>

Risks to participants. Participants on methadone may experience side effects of sedation, constipation, or mild euphoria. The risks of overmedication will be reduced by gradually increasing the dose of methadone over the first week. The methadone dose used in Arm 2 of this protocol, 100 mg, is within the limits allowed by the FDA guidelines and within the dose range used in methadone clinics in Baltimore. For Arm 3 of the protocol, there is no ceiling methadone dose. Methadone doses will be adjusted by the MRP as clinically indicated based on participant feedback, withdrawal signs/symptoms, reported cravings, and urine toxicology results. If a patient shows signs of intoxication, the MRP will reduce the methadone dose until evidence of intoxication has subsided. Methadone will be discontinued if a participant experiences severe side effects. Participants who are withdrawn from methadone will experience opiate withdrawal symptoms, but these symptoms will be minimized by the long detox period of 8 to 12 weeks. Other risks are the inconvenience of carrying and using the EDs, and possible embarrassment from providing urine samples under observation, and concern about the collection of GPS data.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age between 18 and 65;
  2. Evidence of physical dependence on opioids (self-report and physical exam);
  3. Evidence of cocaine and opiate use (self-report and urine screen).

<TAB>

EXCLUSION CRITERIA:

1. Schizophrenia or any other DSM-IV psychotic disorder; history of bipolar disorder; current Major Depressive Disorder;
2. Current dependence on alcohol or sedative-hypnotic, e.g. benzodiazepine (by DSM-IV criteria);
3. Cognitive impairment severe enough to preclude informed consent or valid self-report;
4. Medical illness that in the view of the investigators would compromise participation in research;
5. Urologic conditions that would inhibit urine collection;
6. In arm 2 only: current or recent maintenance on a methadone dose substantially higher than the arm 2 ceiling dose of 100 mg/day; the MRP will evaluate this case by case.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2003-08-15; Study Completion 2013-06-11

CONTACTS AND LOCATIONS:
Overall Officials: Kenzie Preston, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Willner-Reid J, Whitaker D, Epstein DH, Phillips KA, Pulaski AR, Preston KL, Willner P. Cognitive-behavioural therapy for heroin and cocaine use: Ecological momentary assessment of homework simplification and compliance. Psychol Psychother. 2016 Sep;89(3):276-93. doi: 10.1111/papt.12080. Epub 2015 Nov 4. PMID 26530031